CLINICAL TRIAL: NCT03347773
Title: Oral Nutritional Supplement Intervention Among Hemodialysis Patients With Sarcopenic Obesity: a Pilot/Feasibility Randomized Controlled Trial
Brief Title: Oral Nutritional Supplement Intervention Among Hemodialysis Patients With Sarcopenic Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Ting-Yun Lin, Ting-Yun Lin, MD, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 06-M05-079
Record Dates: First submitted 2017-11-12; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Sarcopenic Obesity; Body Composition
Keywords: Oral nutritional supplement; Sarcopenic obesity; Body composition

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The subjects will be assigned to receive nutritional supplement consisting of one can of ReGen 18% (19.1 g protein, 425 Kcal) daily and standard care.
  Interventions: Dietary Supplement: ReGen 18%
- Control (No Intervention): The subjects will be assigned to receive standard care alone.

INTERVENTIONS:
Dietary Supplement: ReGen 18% — ReGen 18% is a kind of oral nutritional supplement, designed for patients under regular hemodialysis. One can of ReGen 18% contains 237ml, 425 Kcal, 19.1g protein, 22.7g lipid and 37.9g carbohydrate.
  Arms: Intervention

SUMMARY:
Chronic kidney disease patients with sarcopenic obesity are noted to have impairment in physical performance and reducing their quality of life, and the investigators also founded these patients are at higher risk of mortality. Thus, the investigators hypothesize that oral nutrition intervention could increase lean tissue mass in these patients and improve the clinical outcomes.

DETAILED DESCRIPTION:
In chronic kidney disease (CKD) patients, disease- and age- related changes in body composition, as well as the increased prevalence of obesity, determine a combination of excess weight and reduced muscle mass or strength, recently defined as sarcopenic obesity. The prevalence of sarcopenic obesity increase with lower eGFR, and previous studies showed that up to 18.3% stage 4 CKD patients and 56% prevalent hemodialysis patient to be with sarcopenic obesity. Sarcopenic obesity was negatively correlated with physical performance and quality of life. In the investigator's previous study, nondialysis-dependent CKD patients with normal body mass index (BMI) but excess body fat had the highest risk of death compared to those with BMI above the cutoff for obesity and excess body fat during a follow up of 5 years. These patients with excess body fat but lower lean tissue mass was what so called "sarcopenic obesity" group.

Hemodialysis therapy per se has been shown to be a catabolic process. Pupim et al. showed that in eight malnourished patients undergoing hemodialysis, highly positive whole-body net protein balance during hemodialysis and improvement of skeletal muscle protein homeostasis was achieved with an intradialytic oral nutritional supplement (ONS) compared to the control, and ONS during hemodialysis resulted in persistent anabolic benefits for muscle protein metabolism in the posthemodialysis phase. In the past, randomized trials of nutritional supplement intervention in dialysis patients were focused on populations with protein energy wasting, and most studies used change in serum albumin concentration as the surrogate marker. Studies focused on dialysis patients with sarcopenic obesity are sparse. Therefore, the investigators hypothesize that ONS could improve the nutritional status among dialysis patients with sarcopenic obesity, especially increase in lean tissue, and improve clinical outcomes. This pilot/feasibility study is aimed to conduct a randomised controlled pilot trial of the feasibility of undertaking a study to assess the effect of ONS on the nutritional status of haemodialysis patients with sarcopenic obesity and will lead to a more robust definitive trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 y/o and 90 y/o
* Regular hemodialysis treatment at least 3 months
* Hemodialysis treatment thrice a week, 3.5-4.5 hours/session
* Body composition: body mass index < 28 kg/m2 and body fat percentage >25% for males or >35% for females
* The normalized protein catabolic rate (nPCR) < 1.2 g/kg/day

Exclusion Criteria:

* Inadequate Kt/V <1.2
* Active malignancy
* Liver cirrhosis
* Active infection, including tuberculosis and AIDS
* Kidney transplant less than 6 months before study enrollment
* Patients hospitalized for more than 5 days within 3 months preceding enrollment
* Patients received intradialytic parental nutrition within 2 months preceding enrollment
* Inability to perform hand grip test, including patients with NG feeding or under bed-ridden status
* Patients with a cardiac pacemaker or metallic implants
* Patients are amputees
* Pregnant woman
* History of poor adherence to dialysis or medication

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in lean tissue mass in kg | Measured at baseline and end of study, 4 months apart
  Measured by bioimpedance device

SECONDARY OUTCOMES:
Change in dry weight in kg | Measured at baseline and end of study, 4 months apart
  Measured by bioimpedance device
Change in body mass index in kg/m^2 | Measured at baseline and end of study, 4 months apart
  Measured by bioimpedance device
Change in fat tissue mass in kg | Measured at baseline and end of study, 4 months apart
  Measured by bioimpedance device
Change in muscle strength in kg | Measured at baseline and end of study, 4 months apart
  Handgrip test
Change in albumin in mg/dl | Measured at baseline and end of study, 4 months apart
  laboratory test
Change in CRP in mg/L. | Measured at baseline and end of study, 4 months apart
  laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yun Lin, MD, Principal Investigator — Taipei Tzu Chi Hospital, Division of Nephrology
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma D, Hawkins M, Abramowitz MK. Association of sarcopenia with eGFR and misclassification of obesity in adults with CKD in the United States. Clin J Am Soc Nephrol. 2014 Dec 5;9(12):2079-88. doi: 10.2215/CJN.02140214. Epub 2014 Nov 12. PMID 25392147
- [Background] Gracia-Iguacel C, Qureshi AR, Avesani CM, Heimburger O, Huang X, Lindholm B, Barany P, Ortiz A, Stenvinkel P, Carrero JJ. Subclinical versus overt obesity in dialysis patients: more than meets the eye. Nephrol Dial Transplant. 2013 Nov;28 Suppl 4:iv175-81. doi: 10.1093/ndt/gft024. PMID 24179011
- [Background] Martinson M, Ikizler TA, Morrell G, Wei G, Almeida N, Marcus RL, Filipowicz R, Greene TH, Beddhu S. Associations of body size and body composition with functional ability and quality of life in hemodialysis patients. Clin J Am Soc Nephrol. 2014 Jun 6;9(6):1082-90. doi: 10.2215/CJN.09200913. Epub 2014 Apr 24. PMID 24763868
- [Background] Pupim LB, Majchrzak KM, Flakoll PJ, Ikizler TA. Intradialytic oral nutrition improves protein homeostasis in chronic hemodialysis patients with deranged nutritional status. J Am Soc Nephrol. 2006 Nov;17(11):3149-57. doi: 10.1681/ASN.2006040413. Epub 2006 Oct 4. PMID 17021267
- [Background] Kalantar-Zadeh K, Cano NJ, Budde K, Chazot C, Kovesdy CP, Mak RH, Mehrotra R, Raj DS, Sehgal AR, Stenvinkel P, Ikizler TA. Diets and enteral supplements for improving outcomes in chronic kidney disease. Nat Rev Nephrol. 2011 May 31;7(7):369-84. doi: 10.1038/nrneph.2011.60. PMID 21629229